CLINICAL TRIAL: NCT05892263
Title: The Study Wonders Whether Early Gastric Force Feeding Can Reduce the Infection Rate and Whether the External Reaction Can Simultaneously Promote the Gastric Motility of the Gastrointestinal Tract Peristalsis Can Reduce the Complications of Postoperative Neck and Wound Anastomosis Leakage, Provide Postoperative Care for Intact Esophagus, and Reduce Postoperative Mortality.
Brief Title: Influence of Early-feeding on Digestive Function of Patients After Esophageal Recontraction Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202205077MIND
Record Dates: First submitted 2022-09-06; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2022-07

CONDITIONS: Early-feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early intestinal force-feeding and drugs to promote gastrointestinal motility (Experimental)
  Interventions: Other: early feeding
- early enteral feeding (Experimental)
  Interventions: Other: early feeding
- giving force-feeding after gas or defecation (No Intervention)

INTERVENTIONS:
Other: early feeding — Enteral force feeding with 5% dextrose injection within 24 hours after operation
  Arms: Early intestinal force-feeding and drugs to promote gastrointestinal motility; early enteral feeding

SUMMARY:
After esophagectomy and reconstruction, intestinal ischemia or intestinal paralysis, lack of intestinal stimulation and oral nutrition can aggravate atrophy and impair the permeability of intestinal mucosa, which not only makes it easy for intestinal bacteria and endotoxin to migrate and enter the blood, At present, early intestinal feeding has been proved to protect the integrity of the intestinal mucosa and improve the postoperative systemic inflammatory response and infection rate of patients, especially pneumonia. Relying on parenteral nutrition, coupled with postoperative exhaust gas or defecation with drugs, can be force-fed. In addition to the side effects of gastrointestinal discomfort (nausea, diarrhea, abdominal pain), parenteral nutrition is likely to cause blood sugar instability and liver index. Abnormal and even increased infection rate, gastrointestinal force feeding was delayed for 36-48 hours before starting.

At present, there is no research on the effect of early force-feeding on gastrointestinal motility. Therefore, this study aims to explore whether early gastrointestinal force-feeding can not only reduce the infection rate and systemic inflammation, but also promote gastrointestinal motility. Without using drugs, Reduce drug side effects and abdominal discomfort, advance the time of gastrointestinal force-feeding, reduce complications of postoperative lung and wound anastomosis leakage, complete postoperative care for esophageal cancer, and reduce postoperative mortality.

At present, there is no research on the effect of early force-feeding on gastrointestinal motility. Therefore, this study aims to explore whether early gastrointestinal force-feeding can not only reduce the infection rate and systemic inflammation, but also promote gastrointestinal motility. Without using drugs, Reduce drug side effects and abdominal discomfort, advance the time of gastrointestinal force-feeding, reduce complications of postoperative lung and wound anastomosis leakage, complete postoperative care for esophageal cancer, and reduce postoperative mortality.

DETAILED DESCRIPTION:
Esophageal rupture, tumor, obstruction, trauma, and dysplasia may all require esophageal reconstruction surgery. Among them, esophageal cancer accounts for the majority. Esophageal cancer is currently one of the most common cancers in the world, and it is also the top six causes of cancer-related deaths. The incidence of esophageal cancer is one of the fastest-growing cancers, and there are obvious differences according to gender and geographical factors. The incidence rate of men is 2-4 times that of women; the incidence rate is the highest in East Asia and southeastern Africa, esophagus The five-year survival rate of cancer is only 5-15%, but the five-year survival rate after surgery can be increased to 40%. Therefore, surgery is currently the preferred treatment for esophageal cancer.

Esophageal cancer surgery is quite complicated, including esophagectomy, radical lymphadenectomy, esophagus and gastric tube re-anastomosis, etc. The difficulty of surgery is related to its high morbidity and mortality. According to the literature review, the overall incidence rate is 59%, and death occurs within 30 days The postoperative complication rate of esophageal cancer is 5%, and the 90-day mortality rate is 13%. Therefore, the treatment of postoperative complications of esophageal cancer is the focus of postoperative care; postoperative complications: shock, pneumonia, anastomotic leakage, delayed gastric emptying, intestinal obstruction, arrhythmia , chylothorax, diaphragmatic hernia, pulmonary embolism, these complications will increase the risk of postoperative death, among which the occurrence of pneumonia leads to a significant increase in mortality and anastomotic leakage as high as 50%.

Radiation therapy before esophagectomy will lead to pulmonary fibrosis, and one-lung ventilation will be used during the operation to increase the surgical field of view for esophageal reconstruction. These two factors lead to a postoperative pulmonary infection rate of 67% in these patients. Unavoidable involvement or sacrifice of the vagus nerve during surgery leads to postoperative complications related to poor digestive function, such as slow gastrointestinal emptying, gastroesophageal reflux, and intestinal obstruction, as high as 39%. The risk of severe pneumonia is a dangerous complication after esophageal surgery; in addition, the esophageal and gastric reconstruction is poorly healed due to gastric juice erosion, resulting in leakage, resulting in systemic sepsis infection and the need for reoperation. It can be seen that gastrointestinal motility after esophageal cancer surgery is related to two common and fatal complications after surgery, which is what needs to be paid more attention to after surgery. If the gastrointestinal function recovers well after surgery, it can be expected to reduce postoperative complications and increase Adequate caloric intake after surgery and accelerated postoperative recovery.

After esophagectomy and reconstruction, intestinal ischemia or intestinal paralysis, lack of intestinal stimulation and oral nutrition can aggravate atrophy and impair the permeability of intestinal mucosa, which not only makes it easy for intestinal bacteria and endotoxin to migrate and enter the blood, At present, early intestinal feeding has been proved to protect the integrity of the intestinal mucosa and improve the postoperative systemic inflammatory response and infection rate of patients, especially pneumonia. Relying on parenteral nutrition, coupled with postoperative exhaust gas or defecation with drugs, can be force-fed. In addition to the side effects of gastrointestinal discomfort (nausea, diarrhea, abdominal pain), parenteral nutrition is likely to cause blood sugar instability and liver index. Abnormal and even increased infection rate, gastrointestinal force feeding was delayed for 36-48 hours before starting.

At present, there is no research on the effect of early force-feeding on gastrointestinal motility. Therefore, this study aims to explore whether early gastrointestinal force-feeding can not only reduce the infection rate and systemic inflammation, but also promote gastrointestinal motility. Without using drugs, Reduce drug side effects and abdominal discomfort, advance the time of gastrointestinal force-feeding, reduce complications of postoperative lung and wound anastomosis leakage, complete postoperative care for esophageal cancer, and reduce postoperative mortality.

ELIGIBILITY:
Inclusion Criteria:

* Esophagectomy
* Esophagectomy ＆ reconstruction
* Esophagotomy
* Esophageal reconstruction-with gastric tube
* Esophageal reconstruction-with colon
* Esophageal reconstruction with small intestine

Exclusion Criteria:

* Gastrointestinal perforation
* Postoperative hemorrhage
* Intestinal obstruction
* Shock

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-07-08 (Estimated); Study Completion 2025-07-08 (Estimated)

PRIMARY OUTCOMES:
gastrointestinal emptying time | up to 24 hours (time of the first bowel movement or exhaust after surgery )
  Start timing the first bowel movement or exhaust time after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No